CLINICAL TRIAL: NCT03424694
Title: HDR Brachytherapy Used as Monotherapy for Low and Intermediate Risk Prostate Cancer: a Phase II Randomized Trial
Brief Title: HDR Brachytherapy as Monotherapy for Low and Intermediate Risk Prostate Cancer
Acronym: BRP2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CR-CSSS Champlain-Charles-Le Moyne (Other)
Responsible Party: Principal Investigator, Marjory Jolicoeur, MD, CR-CSSS Champlain-Charles-Le Moyne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AA-HCLM-14-034
Record Dates: First submitted 2018-01-29; First posted 2018-02-07 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Prostate Cancer
Keywords: Brachytherapy; Monotherapy; HDR Brachytherapy; Toxicity; Quality of Life; Progression Free Survival
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Radiation: HDR brachytherapy monotherapy (1 vs 2 fractions on single implant)
  Brachytherapy in this study consists of treatment with a single interstitial HDR brachytherapy procedures with temporary interstitial catheters. The number of temporary interstitial catheters will be based on the size and shape of the prostate (at least 16 catheters will be implanted).
  In one arm patient will received a single fraction of 19.5 Gray (Gy), in the other arm patient will received 29 Gy/ 2 fractions of 14.5 Gy separated by 6 hours on a single implant.
  Implant will be done with transperineal insertion of interstitial catheters under sterile conditions guided by transrectal ultrasounds.
  Optimization of treatment plan will be done with Oncentra (Elekta) based on MRI imaging done post-implant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2 fractions of 14.5 Gy HDR Brachytherapy (Experimental): High Dose Rate (HDR) Brachytherapy as monotherapy at a dose of 29 Gy is delivered in 2 fractions of 14.5 Gy, minimum 6 hours a part, delivered on a single implant procedure with 2 MRI assisted plannings and dosimetries.
  HDR brachytherapy implant is done under anesthesia with ultrasound guidance as an out-patient procedure.
  Interventions: Radiation: HDR brachytherapy as monotherapy
- 1 fraction of 19.5 Gy HDR brachytherapy (Experimental): HDR Brachytherapy as monotherapy at a dose 19.5 Gy is delivered in 1 fraction. Treatment is done on a single ultrasound guided implant, post implant MRI assisted planning and dosimetry.
  HDR brachytherapy implant is done under anesthesia with ultrasound guidance as an out-patient procedure.
  Interventions: Radiation: HDR brachytherapy as monotherapy

INTERVENTIONS:
Radiation: HDR brachytherapy as monotherapy

SUMMARY:
The purpose of this study is to evaluate High-dose rate (HDR) brachytherapy (1 vs 2 fractions on single implant) as monotherapy for the treatment of low risk and intermediate risk prostate cancer

DETAILED DESCRIPTION:
INTRODUCTION:

Several modalities of radiotherapy treatments are available for low and intermediate risk of prostate cancer, all avec similar results on biochemical control and toxicities. Among them, the brachytherapy consist in the implantation of radioactive sources directly in the prostate. Due to the fast dose shot/application of brachytherapy, the irradiation dose is less damaging to neighbor organs. This specific brachytherapy behavior can enhance the control over cancer while reducing toxicities.

Brachytherapy treatment can be delivered by high-dose-rate (HDR) while, at this time, catheters are implanted in the prostate and retrieved right after treatment (10-15 minutes). HDR brachytherapy dose is more coherent than LDR brachytherapy, because it is not under the risk of loss or migration of its source, neither the variations of prostate size due to swelling or shrinkage after the implantation. A more precise and reproducible dose coverage is accomplished with better preserving of the urethra, bladder, and rectum.

Several authors are investigating HDR brachytherapy and comparing doses and the number of fractions of the different treatment plans.

Morton et al. researched the use of one single fraction of 15 Gray HDR with External Beam Radiation Therapy (EBRT) for the treatment of intermediate risk. The investigators found a progression free survival rate higher than 95% at 5 years follow-up, making this the more used treatment plan at this time.

Since investigators already have good control rates with LDR brachytherapy for low and intermediate risk cancers with lower toxicity rates, investigators began to question the need of adjunct external radiotherapy. Besides those rates, HDR brachytherapy has other advantages such as: Medical staff is not subjected to radiation, no radiation source is left on the patient's body, treatment time is decreased from several months to few minutes, and the dose distribution is better used because of the capacity to precisely control the source position during treatment.

HDR brachytherapy is usually given is small fraction number, but the optimal fraction number for HDR monotherapy is unknown. Most researchers prescribe 4 to 6 fractions, with a 6 hours interval between fractions. Catheters are left in place and treatment lasts from two to several days, unavoidably needing patient's hospitalisation. Another possible inconvenience is the possible catheters displacement between fractions, leading to verifications and corrections before each fraction is delivered. Trying to reduce the number of fractions and give enough dose is being studied in several institutions. The dose is not only related to the efficacy of the treatment, but also to the toxicities related to it.

The purpose of this study is to evaluate High-dose rate (HDR) brachytherapy (1 vs 2 fractions on single implant) as monotherapy for the treatment of low risk and intermediate risk prostate cancer. One fraction HDR brachytherapy will be delivered in one 19.5 Gy dose, while the two fractions will be delivered in two fractions of 14.5 Gy (total dose of 29Gy), both on single implant procedure. This evaluation will be carried under a single institution as a phase II randomized clinical trial (RTC) design.

Hypothesis:

The HDR brachytherapy as monotherapy given in one or two fractions (one fraction of 19.5 Gy or two fractions of 14.5Gy) is well tolerated and effective for the treatment of low and intermediate risk prostate cancers.

Objectives:

Primary Objective:

The aim of this study is to evaluate acute (early) toxicities (genitourinary and gastrointestinal) of HDR brachytherapy (1 vs 2 fractions on single implant) as monotherapy for low and intermediate risk prostate cancer.

Secondary Objectives:

* Measure overall survival and progression free survival rate
* Evaluate the evolution of the International Prostate Symptom Score (IPSS) and its time to return to baseline.
* Evaluate late genitourinary and gastrointestinal toxicities changes measured by RTOG and CTCAE v4 score
* Evaluate biochemical failure
* Evaluate erectile dysfunction rates
* Investigate associations between dosimetric parameters and toxicity
* Investigate associations between iUrethra parameters and toxicity
* Assess changes in the quality of life of patients - EORTC QLQ-C30

METHODS:

Patient's selection and randomization:

Inclusion and exclusion criteria are described elsewhere. Once patients fullfil all selection criteria they will be randomized between one of the 2 arms of the study (1 or 2 fractions) by sealed envelope system.

Treatment:

Patients will undergo preoperative standard care conditions. The procedure will be taken under regional anesthesia with sterile conditions; Foley urinary catheter will be inserted and will aid the urethra delimitation. The bladder will be emptied and the catheter will be clamped. Transrectal ultrasound (TRUS) will guide the placement of the transperineal catheters. The number of temporary interstitial catheters will be based on the size and shape of the prostate (at least 16 catheters will be implanted).

Optimization of treatment plan will be done with Oncentra (Elekta) based on MRI imaging done post-implant. The following contours will be delimited: the prostate, the urinary catheter (urethra), the urethra as seen on the MRI (iUrethra), the rectum and the bladder. Catheters will be rebuilt on the planning system. The dose calculations will be done by reverse planning. After treatment, catheters will be removed and the patient will be transferred to the recovery room. Patient will be sent home after recovery with urinary catheter. Urinary catheter will be retrieved the day after.

Patients receiving two fractions will undergo CT scan before the second fraction, if the catheters have to be repositioned, appropriate adjustments will be made to optimize the dose distribution and correct any changes in dosimetry of the implant.

Patient's evaluation:

After the end of treatment, patients will be seen at 1, 3 and 6 weeks, 3 months, 6 months, 12 months and then every 6 months until year 5. PSA, IPSS, IIEF5 and EORTC QLQ-C30 will be fulfilled during follow-up appointments.

Procedures for biochemical recurrence will be at the discretion of the attending physician.

New biopsies will not be performed if local recurrence is suspected and that the metastatic work-up (abdominopelvic CT scan, bone scintigraphy) is positive. Nevertheless, in cases of suspicion of local or remote recccurence investigation will take place.

Statistics:

The assumption is that for each arm the probability of a standard deviation difference will be higher than 0.5 of the urinary toxicities at one year compared to the baseline will be lower than or equal to our current standards.

Sample size:

To detect this difference, the test of proportions was used with the NCSS / PASS software. The sample size was estimated at 180 patients (90 per arm) calculated with 99% power and a 0.05 significance level (one-tail test). Considering 10% ineligibility, the required sample size is 200 patients (100 per arm).

Statistical analysis:

Statistical analysis will be performed at SAS 9.3 software package. Anova repeated measures (Mixed Models) and regression logistic regression models (GEE: Generalized Estimation Equations) will be used.

These multivariate models will allow us to determine the potential associations between our dependent variables while controlling as much for socio-demographic factors and especially for potentially confounding clinical variables.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven prostate adenocarcinoma
* Clinical Stage T1c - T2c
* Gleason Score between 6 and 7
* PSA < 15 ng / ml
* Prostate volume < 70 cc as determined by ultrasound or IRM
* Signed informer consent
* Clinical conditions for complete diagnosis checkup and treatment procedure
* Should be able to complete IIEFS,IPSS and QLQ-C30 questionnaires
* Bone and pelvic scan negative for metastasis

Exclusion Criteria:

* Prior pelvis radiation
* Prior Transurethral resection of the prostate (TURP) (less than 6 months)
* International Prostate Symptom Score: IPSS > 16
* Contraindication to radiotherapy
* No prior use of Androgen deprivation therapy (ADT)
* Observation: 5 alpha-reductase (5AR) inhibitors is authorized.

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 199 (Actual)
Dates: Start 2015-06-22 (Actual); Primary Completion 2019-06-22 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
Acute (early) genitourinary and gastrointestinal toxicity | 10 years
  Acute genitourinary and gastrointestinal toxicities of HDR Brachytherapy will be graded using the Radiation Therapy Oncology Group (RTOG) Score at each follow up time point.

SECONDARY OUTCOMES:
Overall survival | 10 years
  The difference in median overall survival will be compared between the two arms.
  Overall survival (OS) measured in months from baseline to death from any cause.
Local - Progression free survival (PFS) | 10 years
  The difference in median PFS will be compared between the two arms. Progression free survival (PFS) measured in months from baseline to local disease relapse.
Distant - Progression free survival (PFS) | 10 years
  The difference in median PFS will be compared between the two arms. Progression free survival (PFS) measured in months from baseline to distant disease relapse.
Evolution of the International Prostate Symptom Score (IPSS) and time to return to baseline | 3 years
  IPSS scores will be measured at baseline, 1 week, 3 weeks, 6 weeks, 6 months, 12 months, 24 months and 36 months.
Late genitourinary and gastrointestinal toxicities changes | 10 years
  Late Late genitourinary and gastrointestinal toxicities measured measured by CTCAE v4 and RTOG score
Biochemical failure | 10 years
  PSA measure changes will be recorded every 3 months for the first 2 years, every 6 months to 5 years and then annually to 10 years.
Erectile dysfunction rates - IIEF5 score | 3 years
  IIEF5 scores will be measured at baseline, 1 week, 3 weeks, 6 weeks, 6 months, 12 months, 24 months and 36 months.
Associations between dosimetric parameters and toxicity | 3 years
  Patients with symptomatic prostatitis will be identified
Associations between iUrethra and toxicity | 3 years
  iUrethra is represented by urethra MRI imaging and draw upon the length of the previous targeted volume (1cm inferior and superior margins).
  iUrethra differs from the urethra measure, since it is not draw upon the urinary catheter.
Changes in the quality of life of patients - EORTC QLQ-C30 | 5 years
  Scores will be evaluated at baseline, 1, 3, 6, 12, 24, 36 and 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Marjory Jolicoeur, MD, Principal Investigator — CSSS Champlain-Charles-Le Moyne
Locations (1):
- Hôpital Charles LeMoyne, Greenfield Park, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang Y, Sankreacha R, Al-Hebshi A, Loblaw A, Morton G. Comparative study of dosimetry between high-dose-rate and permanent prostate implant brachytherapies in patients with prostate adenocarcinoma. Brachytherapy. 2006 Oct-Dec;5(4):251-5. doi: 10.1016/j.brachy.2006.08.006. PMID 17118319
- [Background] Davis BJ, Horwitz EM, Lee WR, Crook JM, Stock RG, Merrick GS, Butler WM, Grimm PD, Stone NN, Potters L, Zietman AL, Zelefsky MJ; American Brachytherapy Society. American Brachytherapy Society consensus guidelines for transrectal ultrasound-guided permanent prostate brachytherapy. Brachytherapy. 2012 Jan-Feb;11(1):6-19. doi: 10.1016/j.brachy.2011.07.005. PMID 22265434
- [Background] Herbert C, Morris WJ, Keyes M, Hamm J, Lapointe V, McKenzie M, Pickles T, Spadinger I. Outcomes following iodine-125 brachytherapy in patients with Gleason 7, intermediate risk prostate cancer: a population-based cohort study. Radiother Oncol. 2012 May;103(2):228-32. doi: 10.1016/j.radonc.2012.01.006. Epub 2012 Feb 10. PMID 22326573
- [Background] Morton GC. The emerging role of high-dose-rate brachytherapy for prostate cancer. Clin Oncol (R Coll Radiol). 2005 Jun;17(4):219-27. doi: 10.1016/j.clon.2004.12.005. PMID 15997914
- [Background] Yamada Y, Rogers L, Demanes DJ, Morton G, Prestidge BR, Pouliot J, Cohen GN, Zaider M, Ghilezan M, Hsu IC; American Brachytherapy Society. American Brachytherapy Society consensus guidelines for high-dose-rate prostate brachytherapy. Brachytherapy. 2012 Jan-Feb;11(1):20-32. doi: 10.1016/j.brachy.2011.09.008. PMID 22265435
- [Background] Bachand F, Martin AG, Beaulieu L, Harel F, Vigneault E. An eight-year experience of HDR brachytherapy boost for localized prostate cancer: biopsy and PSA outcome. Int J Radiat Oncol Biol Phys. 2009 Mar 1;73(3):679-84. doi: 10.1016/j.ijrobp.2008.05.003. Epub 2008 Oct 27. PMID 18963537
- [Background] Martinez AA, Gonzalez J, Ye H, Ghilezan M, Shetty S, Kernen K, Gustafson G, Krauss D, Vicini F, Kestin L. Dose escalation improves cancer-related events at 10 years for intermediate- and high-risk prostate cancer patients treated with hypofractionated high-dose-rate boost and external beam radiotherapy. Int J Radiat Oncol Biol Phys. 2011 Feb 1;79(2):363-70. doi: 10.1016/j.ijrobp.2009.10.035. PMID 21195875
- [Background] Deutsch I, Zelefsky MJ, Zhang Z, Mo Q, Zaider M, Cohen G, Cahlon O, Yamada Y. Comparison of PSA relapse-free survival in patients treated with ultra-high-dose IMRT versus combination HDR brachytherapy and IMRT. Brachytherapy. 2010 Oct-Dec;9(4):313-8. doi: 10.1016/j.brachy.2010.02.196. Epub 2010 Aug 4. PMID 20685176
- [Background] Hoskin PJ, Rojas AM, Bownes PJ, Lowe GJ, Ostler PJ, Bryant L. Randomised trial of external beam radiotherapy alone or combined with high-dose-rate brachytherapy boost for localised prostate cancer. Radiother Oncol. 2012 May;103(2):217-22. doi: 10.1016/j.radonc.2012.01.007. Epub 2012 Feb 16. PMID 22341794
- [Background] Morton GC, Loblaw DA, Sankreacha R, Deabreu A, Zhang L, Mamedov A, Cheung P, Keller B, Danjoux C, Szumacher E, Thomas G. Single-fraction high-dose-rate brachytherapy and hypofractionated external beam radiotherapy for men with intermediate-risk prostate cancer: analysis of short- and medium-term toxicity and quality of life. Int J Radiat Oncol Biol Phys. 2010 Jul 1;77(3):811-7. doi: 10.1016/j.ijrobp.2009.05.054. Epub 2009 Oct 14. PMID 19836166
- [Background] Cury FL, Duclos M, Aprikian A, Patrocinio H, Kassouf W, Shenouda G, Faria S, David M, Souhami L. Single-fraction high-dose-rate brachytherapy and hypofractionated external beam radiation therapy in the treatment of intermediate-risk prostate cancer - long term results. Int J Radiat Oncol Biol Phys. 2012 Mar 15;82(4):1417-23. doi: 10.1016/j.ijrobp.2011.05.025. Epub 2011 Jul 23. PMID 21784585
- [Background] Morton G, Loblaw A, Cheung P, Szumacher E, Chahal M, Danjoux C, Chung HT, Deabreu A, Mamedov A, Zhang L, Sankreacha R, Vigneault E, Springer C. Is single fraction 15 Gy the preferred high dose-rate brachytherapy boost dose for prostate cancer? Radiother Oncol. 2011 Sep;100(3):463-7. doi: 10.1016/j.radonc.2011.08.022. Epub 2011 Sep 14. PMID 21924511
- [Background] Taira AV, Merrick GS, Galbreath RW, Wallner KE, Butler WM. Natural history of clinically staged low- and intermediate-risk prostate cancer treated with monotherapeutic permanent interstitial brachytherapy. Int J Radiat Oncol Biol Phys. 2010 Feb 1;76(2):349-54. doi: 10.1016/j.ijrobp.2009.02.021. Epub 2009 May 19. PMID 19467793
- [Background] Barkati M, Williams SG, Foroudi F, Tai KH, Chander S, van Dyk S, See A, Duchesne GM. High-dose-rate brachytherapy as a monotherapy for favorable-risk prostate cancer: a Phase II trial. Int J Radiat Oncol Biol Phys. 2012 Apr 1;82(5):1889-96. doi: 10.1016/j.ijrobp.2010.09.006. Epub 2011 May 6. PMID 21550182
- [Background] Demanes DJ, Martinez AA, Ghilezan M, Hill DR, Schour L, Brandt D, Gustafson G. High-dose-rate monotherapy: safe and effective brachytherapy for patients with localized prostate cancer. Int J Radiat Oncol Biol Phys. 2011 Dec 1;81(5):1286-92. doi: 10.1016/j.ijrobp.2010.10.015. Epub 2011 Feb 9. PMID 21310546
- [Background] Rogers CL, Alder SC, Rogers RL, Hopkins SA, Platt ML, Childs LC, Crouch RH, Hansen RS, Hayes JK. High dose brachytherapy as monotherapy for intermediate risk prostate cancer. J Urol. 2012 Jan;187(1):109-16. doi: 10.1016/j.juro.2011.09.050. Epub 2011 Nov 16. PMID 22088340
- [Background] Martinez AA, Demanes J, Vargas C, Schour L, Ghilezan M, Gustafson GS. High-dose-rate prostate brachytherapy: an excellent accelerated-hypofractionated treatment for favorable prostate cancer. Am J Clin Oncol. 2010 Oct;33(5):481-8. doi: 10.1097/COC.0b013e3181b9cd2f. PMID 19952715
- [Background] Holly R, Morton GC, Sankreacha R, Law N, Cisecki T, Loblaw DA, Chung HT. Use of cone-beam imaging to correct for catheter displacement in high dose-rate prostate brachytherapy. Brachytherapy. 2011 Jul-Aug;10(4):299-305. doi: 10.1016/j.brachy.2010.11.007. Epub 2010 Dec 28. PMID 21190903
- [Background] Kolkman-Deurloo IK, Roos MA, Aluwini S. HDR monotherapy for prostate cancer: a simulation study to determine the effect of catheter displacement on target coverage and normal tissue irradiation. Radiother Oncol. 2011 Feb;98(2):192-7. doi: 10.1016/j.radonc.2010.12.009. Epub 2011 Feb 3. PMID 21295878
- [Background] Ghilezan M, Martinez A, Gustason G, Krauss D, Antonucci JV, Chen P, Fontanesi J, Wallace M, Ye H, Casey A, Sebastian E, Kim L, Limbacher A. High-dose-rate brachytherapy as monotherapy delivered in two fractions within one day for favorable/intermediate-risk prostate cancer: preliminary toxicity data. Int J Radiat Oncol Biol Phys. 2012 Jul 1;83(3):927-32. doi: 10.1016/j.ijrobp.2011.05.001. Epub 2011 Dec 23. PMID 22197086
- [Background] Hoskin P, Rojas A, Lowe G, Bryant L, Ostler P, Hughes R, Milner J, Cladd H. High-dose-rate brachytherapy alone for localized prostate cancer in patients at moderate or high risk of biochemical recurrence. Int J Radiat Oncol Biol Phys. 2012 Mar 15;82(4):1376-84. doi: 10.1016/j.ijrobp.2011.04.031. Epub 2011 Jun 15. PMID 21680108
- [Background] Prada PJ, Jimenez I, Gonzalez-Suarez H, Fernandez J, Cuervo-Arango C, Mendez L. High-dose-rate interstitial brachytherapy as monotherapy in one fraction and transperineal hyaluronic acid injection into the perirectal fat for the treatment of favorable stage prostate cancer: treatment description and preliminary results. Brachytherapy. 2012 Mar-Apr;11(2):105-10. doi: 10.1016/j.brachy.2011.05.003. Epub 2011 Sep 14. PMID 21917528
- [Background] Morton GC, Loblaw DA, Chung H, Tsang G, Sankreacha R, Deabreu A, Zhang L, Mamedov A, Cheung P, Batchelar D, Danjoux C, Szumacher E. Health-related quality of life after single-fraction high-dose-rate brachytherapy and hypofractionated external beam radiotherapy for prostate cancer. Int J Radiat Oncol Biol Phys. 2011 Aug 1;80(5):1299-305. doi: 10.1016/j.ijrobp.2010.04.046. Epub 2010 Aug 12. PMID 20708853
- [Background] Yoshioka Y, Konishi K, Oh RJ, Sumida I, Yamazaki H, Nakamura S, Nishimura K, Nonomura N, Okuyama A, Inoue T. High-dose-rate brachytherapy without external beam irradiation for locally advanced prostate cancer. Radiother Oncol. 2006 Jul;80(1):62-8. doi: 10.1016/j.radonc.2006.06.011. Epub 2006 Jul 25. PMID 16870289
- [Background] Hoskin P, Rojas A, Ostler P, Hughes R, Alonzi R, Lowe G, Bryant L. High-dose-rate brachytherapy alone given as two or one fraction to patients for locally advanced prostate cancer: acute toxicity. Radiother Oncol. 2014 Feb;110(2):268-71. doi: 10.1016/j.radonc.2013.09.025. Epub 2013 Nov 11. PMID 24231242
- [Background] Jolicoeur, M., Derashodian, T., Last, J., Wakil, G., & Mondat, M. (2017). Multimodality Image Registrations for Combined MRI/CT HDR Prostate Brachytherapy: The Concept of the Iurethra. International Journal of Radiation Oncology*Biology*Physics, 99(2), E243-E244. https://doi.org/10.1016/J.IJROBP.2017.06.1185